CLINICAL TRIAL: NCT02704156
Title: Stereotactic Body Radiation Therapy Plus Pembrolizumab and Trametinib vs. Stereotactic Body Radiation Therapy Plus Gemcitabine for Locally Recurrent Pancreatic Cancer After Surgical Resection: an Open-label, Randomized, Controlled, Phase 2 Trial
Brief Title: SBRT Plus Pembrolizumab and Trametinib for Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhang Huo Jun, Director of Radiation Oncology Department, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChanghaiHosp
Record Dates: First submitted 2016-03-01; First posted 2016-03-09 (Estimated); Results first posted 2021-02-16 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-02

CONDITIONS: Pancreatic Cancer
Keywords: Stereotactic body radiation therapy; CyberKnife; Initial treatment
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SBRT plus Pembrolizumab and Trametinib (Experimental): Patients with locally recurrent pancreatic cancer were randomly allocated to SBRT plus Pembrolizumab and Trametinib or SBRT plus Gemcitabine.
  Interventions: Device: Cyberknife plus Pembrolizumab and Trametinib
- SBRT plus Gemcitabine (Active Comparator): Patients with locally recurrent pancreatic cancer were randomly allocated to SBRT plus Pembrolizumab and Trametinib or SBRT plus Gemcitabine.
  Interventions: Device: Cyberknife plus Gemcitabine

INTERVENTIONS:
Device: Cyberknife plus Pembrolizumab and Trametinib — Radiation therapy plus drug
  Arms: SBRT plus Pembrolizumab and Trametinib
Device: Cyberknife plus Gemcitabine — Radiation therapy plus drug
  Arms: SBRT plus Gemcitabine

SUMMARY:
Hypothesis: Survival benefits could be found in SBRT Plus Pembrolizumab and Trametinib compared with SBRT plus gemcitabine.

DETAILED DESCRIPTION:
Background and aim:

Pancreatic cancer is one of the most lethal malignancies and fourth leading cause of cancer death in both genders in US, where the mortality and incidence increase over the past decade with a lowest 5-year survival rate of 9% among all cancers. Although surgical resection is deemed to provide long-term disease control, only 20% patients were candidates for upfront surgery and unfortunately, even when adjuvant chemotherapy is prescribed, about 50% of patients will suffer local recurrence. Despite of emergence of immunotherapy as a new treatment paradigm, little improvement of outcomes has been found in pancreatic cancer. This may be ascribed to its inherent genetic mutations and immunosuppressive microenvironment. It has been demonstrated that radiotherapy could enhance the release and uptake of tumor-associated antigens, thus promoting antitumor T cell priming, and enhancing access to tumors due to effects both on the tumor vasculature and the chemokine milieu.

Despite of emergence of immune checkpoint inhibitors as a novel treatment paradigm for cancers, the results of investigations about the efficacy of immunotherapy alone for pancreatic cancer was disappointing. Due to enhanced immunogenicity of tumor irradiation, the underlying rationale of combination of radiotherapy and immunotherapy is that radiation can noninvasively prime the immune system against tumor cells, where antigen presentation and co-stimulation are facilitated, thus creating immune responses against previously hidden epitopes that are shared among distant metastases, while immune checkpoint inhibitors can reverse the immunosuppressive effects of the tumor microenvironment, thus facilitating antitumor immunity.

Although oncogenic mutations in KRAS are frequent in pancreatic cancer, KRAS proteins are difficult to be targeted due to high affinity for GTP and/or GDP. Therefore, efforts have been made to develop therapies targeting the major downstream effector pathways, which include the RAS-RAF-MEK-ERK and PI3K-PDPK1-AKT signaling pathways. MEK inhibitor trametinib alone or in combinations with chemotherapy or autophagy inhibitor hydroxychloroquine may probably have positive effects on tumor regression.

Regarding local recurrence after surgery, it was recommended that chemotherapy with optional radiotherapy may be the first-line treatment without addition of targeted therapy or immunotherapy owing to that no studies have investigated the efficacy of this regimen. Therefore, the aim of our study was to compare the outcomes between stereotactic body radiation therapy (SBRT) with pembrolizumab and trametinib and SBRT with gemcitabine for locally recurrent pancreatic cancer after surgical resection.

Study procedure:

1. All surgical specimens underwent immunohistochemical staining of PD-L1, classified as TC3 ≥ 50% or TC2 ≥ 5% but < 50% or TC1 ≥ 1% but <5% and IC3 ≥ 10% or IC2 ≥ 5% but < 10% or IC1 ≥ 1% but <5%.
2. KRAS mutations were analyzed by PCR amplification and direct sequencing of exon 2. Restriction Length Fragment Polymorphism method was used for further confirmation.
3. In the SBRT plus pembrolizumab and trametinib group, 200mg pembrolizumab was administered intravenously every 3 weeks and 2mg trametinib was given orally once daily.
4. In the SBRT plus gemcitabine group, patients received intravenous gemcitabine (1000mg/m2) on day 1 and 8 of each 21-day cycle for eight cycles in the absence of disease progression.
5. The prescribed dose of SBRT varies from 35-40Gy/5f with a single dose of 7-8Gy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed pancreatic ductal adenocarcinoma with unequivocal first progression after surgery followed by chemotherapy
2. Without any immunotherapy or targeted therapy
3. A life expectancy of >3months
4. ECOG of 0 to1
5. Age of 18 years or older
6. Analysis of surgical specimens showed KRAS mutations and positive immunohistochemical staining of PD-L1
7. Blood routine examination: Absolute neutrophil count (ANC) ≥ 1.5 ×109 cells/L, leukocyte count≥ 3.5 ×109 cells/L, platelets ≥ 70×109 cells/L, hemoglobin ≥ 8.0 g/dl
8. Liver and kidney function tests: Albumin > 2.5 g/dL, total bilirubin < 3 mg/dL, creatinine < 2.0 mg/dL, AST<2.5 × ULN(Upper Limit of Normal)(0-64U/L), ALT<2.5 × ULN(0-64U/L)
9. INR < 2 (0.9-1.1)
10. Ability of the research subject or authorized legal representative to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Prior immunotherapy or targeted therapy
2. Evidences of metastatic disease confirmed by chest CT or FDG PET-CT
3. Contraindication to receiving immunotherapy, targeted therapy or SBRT
4. ECOG ≥2
5. Age <18 years
6. Analysis of surgical specimens showed KRAS wild type or negative immunohistochemical staining of PD-L1
7. Secondary malignancy
8. Abnormal results of blood routine examinations and liver and kidney and coagulation tests
9. Patients with active inflammatory bowel diseases or peptic ulcer
10. Gastrointestinal bleeding or perforation within 6 months
11. Heart failure: NYHA III-IV
12. Respiratory insufficiency
13. Women who are pregnant
14. Participation in another clinical treatment trial while on study
15. Patients in whom fiducial implantation was not possible
16. Inability of the research subject or authorized legal representative to understand and the willingness to sign a written informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huo Jun Zhang, MD., PH.D, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Siegel RL, Miller KD, Goding Sauer A, Fedewa SA, Butterly LF, Anderson JC, Cercek A, Smith RA, Jemal A. Colorectal cancer statistics, 2020. CA Cancer J Clin. 2020 May;70(3):145-164. doi: 10.3322/caac.21601. Epub 2020 Mar 5. PMID 32133645
- [Background] Oettle H, Neuhaus P, Hochhaus A, Hartmann JT, Gellert K, Ridwelski K, Niedergethmann M, Zulke C, Fahlke J, Arning MB, Sinn M, Hinke A, Riess H. Adjuvant chemotherapy with gemcitabine and long-term outcomes among patients with resected pancreatic cancer: the CONKO-001 randomized trial. JAMA. 2013 Oct 9;310(14):1473-81. doi: 10.1001/jama.2013.279201. PMID 24104372
- [Background] Dewan MZ, Galloway AE, Kawashima N, Dewyngaert JK, Babb JS, Formenti SC, Demaria S. Fractionated but not single-dose radiotherapy induces an immune-mediated abscopal effect when combined with anti-CTLA-4 antibody. Clin Cancer Res. 2009 Sep 1;15(17):5379-88. doi: 10.1158/1078-0432.CCR-09-0265. Epub 2009 Aug 25. PMID 19706802
- [Background] Verbrugge I, Hagekyriakou J, Sharp LL, Galli M, West A, McLaughlin NM, Duret H, Yagita H, Johnstone RW, Smyth MJ, Haynes NM. Radiotherapy increases the permissiveness of established mammary tumors to rejection by immunomodulatory antibodies. Cancer Res. 2012 Jul 1;72(13):3163-74. doi: 10.1158/0008-5472.CAN-12-0210. Epub 2012 May 8. PMID 22570253
- [Background] Royal RE, Levy C, Turner K, Mathur A, Hughes M, Kammula US, Sherry RM, Topalian SL, Yang JC, Lowy I, Rosenberg SA. Phase 2 trial of single agent Ipilimumab (anti-CTLA-4) for locally advanced or metastatic pancreatic adenocarcinoma. J Immunother. 2010 Oct;33(8):828-33. doi: 10.1097/CJI.0b013e3181eec14c. PMID 20842054
- [Background] Brahmer JR, Tykodi SS, Chow LQ, Hwu WJ, Topalian SL, Hwu P, Drake CG, Camacho LH, Kauh J, Odunsi K, Pitot HC, Hamid O, Bhatia S, Martins R, Eaton K, Chen S, Salay TM, Alaparthy S, Grosso JF, Korman AJ, Parker SM, Agrawal S, Goldberg SM, Pardoll DM, Gupta A, Wigginton JM. Safety and activity of anti-PD-L1 antibody in patients with advanced cancer. N Engl J Med. 2012 Jun 28;366(26):2455-65. doi: 10.1056/NEJMoa1200694. Epub 2012 Jun 2. PMID 22658128
- [Background] Chakraborty M, Abrams SI, Coleman CN, Camphausen K, Schlom J, Hodge JW. External beam radiation of tumors alters phenotype of tumor cells to render them susceptible to vaccine-mediated T-cell killing. Cancer Res. 2004 Jun 15;64(12):4328-37. doi: 10.1158/0008-5472.CAN-04-0073. PMID 15205348
- [Background] Bailey P, Chang DK, Nones K, Johns AL, Patch AM, Gingras MC, Miller DK, Christ AN, Bruxner TJ, Quinn MC, Nourse C, Murtaugh LC, Harliwong I, Idrisoglu S, Manning S, Nourbakhsh E, Wani S, Fink L, Holmes O, Chin V, Anderson MJ, Kazakoff S, Leonard C, Newell F, Waddell N, Wood S, Xu Q, Wilson PJ, Cloonan N, Kassahn KS, Taylor D, Quek K, Robertson A, Pantano L, Mincarelli L, Sanchez LN, Evers L, Wu J, Pinese M, Cowley MJ, Jones MD, Colvin EK, Nagrial AM, Humphrey ES, Chantrill LA, Mawson A, Humphris J, Chou A, Pajic M, Scarlett CJ, Pinho AV, Giry-Laterriere M, Rooman I, Samra JS, Kench JG, Lovell JA, Merrett ND, Toon CW, Epari K, Nguyen NQ, Barbour A, Zeps N, Moran-Jones K, Jamieson NB, Graham JS, Duthie F, Oien K, Hair J, Grutzmann R, Maitra A, Iacobuzio-Donahue CA, Wolfgang CL, Morgan RA, Lawlor RT, Corbo V, Bassi C, Rusev B, Capelli P, Salvia R, Tortora G, Mukhopadhyay D, Petersen GM; Australian Pancreatic Cancer Genome Initiative; Munzy DM, Fisher WE, Karim SA, Eshleman JR, Hruban RH, Pilarsky C, Morton JP, Sansom OJ, Scarpa A, Musgrove EA, Bailey UM, Hofmann O, Sutherland RL, Wheeler DA, Gill AJ, Gibbs RA, Pearson JV, Waddell N, Biankin AV, Grimmond SM. Genomic analyses identify molecular subtypes of pancreatic cancer. Nature. 2016 Mar 3;531(7592):47-52. doi: 10.1038/nature16965. Epub 2016 Feb 24. PMID 26909576
- [Background] McCormick F. KRAS as a Therapeutic Target. Clin Cancer Res. 2015 Apr 15;21(8):1797-801. doi: 10.1158/1078-0432.CCR-14-2662. PMID 25878360
- [Background] Eser S, Schnieke A, Schneider G, Saur D. Oncogenic KRAS signalling in pancreatic cancer. Br J Cancer. 2014 Aug 26;111(5):817-22. doi: 10.1038/bjc.2014.215. Epub 2014 Apr 22. PMID 24755884
- [Background] Vena F, Li Causi E, Rodriguez-Justo M, Goodstal S, Hagemann T, Hartley JA, Hochhauser D. The MEK1/2 Inhibitor Pimasertib Enhances Gemcitabine Efficacy in Pancreatic Cancer Models by Altering Ribonucleotide Reductase Subunit-1 (RRM1). Clin Cancer Res. 2015 Dec 15;21(24):5563-77. doi: 10.1158/1078-0432.CCR-15-0485. Epub 2015 Jul 30. PMID 26228206
- [Background] Kinsey CG, Camolotto SA, Boespflug AM, Guillen KP, Foth M, Truong A, Schuman SS, Shea JE, Seipp MT, Yap JT, Burrell LD, Lum DH, Whisenant JR, Gilcrease GW 3rd, Cavalieri CC, Rehbein KM, Cutler SL, Affolter KE, Welm AL, Welm BE, Scaife CL, Snyder EL, McMahon M. Protective autophagy elicited by RAF-->MEK-->ERK inhibition suggests a treatment strategy for RAS-driven cancers. Nat Med. 2019 Apr;25(4):620-627. doi: 10.1038/s41591-019-0367-9. Epub 2019 Mar 4. PMID 30833748
- [Background] Bryant KL, Stalnecker CA, Zeitouni D, Klomp JE, Peng S, Tikunov AP, Gunda V, Pierobon M, Waters AM, George SD, Tomar G, Papke B, Hobbs GA, Yan L, Hayes TK, Diehl JN, Goode GD, Chaika NV, Wang Y, Zhang GF, Witkiewicz AK, Knudsen ES, Petricoin EF 3rd, Singh PK, Macdonald JM, Tran NL, Lyssiotis CA, Ying H, Kimmelman AC, Cox AD, Der CJ. Combination of ERK and autophagy inhibition as a treatment approach for pancreatic cancer. Nat Med. 2019 Apr;25(4):628-640. doi: 10.1038/s41591-019-0368-8. Epub 2019 Mar 4. PMID 30833752
- [Derived] Zhu X, Liu W, Cao Y, Ju X, Zhao X, Jiang L, Ye Y, Zhang H. Effect of stereotactic body radiotherapy dose escalation plus pembrolizumab and trametinib versus stereotactic body radiotherapy dose escalation plus gemcitabine for locally recurrent pancreatic cancer after surgical resection on survival outcomes: A secondary analysis of an open-label, randomised, controlled, phase 2 trial. EClinicalMedicine. 2022 Dec 1;55:101764. doi: 10.1016/j.eclinm.2022.101764. eCollection 2023 Jan. PMID 36471691
- [Derived] Zhu X, Cao Y, Liu W, Ju X, Zhao X, Jiang L, Ye Y, Jin G, Zhang H. Stereotactic body radiotherapy plus pembrolizumab and trametinib versus stereotactic body radiotherapy plus gemcitabine for locally recurrent pancreatic cancer after surgical resection: an open-label, randomised, controlled, phase 2 trial. Lancet Oncol. 2022 Mar;23(3):e105-e115. doi: 10.1016/S1470-2045(22)00066-3. PMID 35240087
- [Derived] Zhu X, Cao Y, Liu W, Ju X, Zhao X, Jiang L, Ye Y, Jin G, Zhang H. Stereotactic body radiotherapy plus pembrolizumab and trametinib versus stereotactic body radiotherapy plus gemcitabine for locally recurrent pancreatic cancer after surgical resection: an open-label, randomised, controlled, phase 2 trial. Lancet Oncol. 2021 Aug;22(8):1093-1102. doi: 10.1016/S1470-2045(21)00286-2. Epub 2021 Jul 5. PMID 34237249

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment date was from October 2016 to October 2017. Patients were enrolled in our center.
Period: Overall Study
Arm/Group | SBRT Plus Gemcitabine | SBRT Plus Pembrolizumab and Trametinib
Started | 85 | 85
Completed | 85 | 85
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SBRT Plus Gemcitabine | SBRT Plus Pembrolizumab and Trametinib | Total
Number analyzed (Participants) | 85 | 85 | 170
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [58 to 73] | 65 [54 to 74] | 65 [57 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 32 | 65
  Male | 52 | 53 | 105
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 85 | 85 | 170
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 85 | 85 | 170
PD-L1 intensity [Number; unit: participants] — PD-L1 tumor cell (TC) expression was scored as the percentage of PD-L1 TC, which was stratified as TC3 ≥ 50% or TC2 ≥ 5% but < 50% or TC1 ≥ 1% but <5%. PD-L1 tumor-infiltrating immune cells (IC) expression was scored as the percentage of tumor area stained positive, which was classified as IC3 ≥ 10% or IC2 ≥ 5% but < 10% or IC1 ≥ 1% but <5%. Briefly, the higher expression of TCor IC indicated worse outcomes.
  participants
    IC1 or TC1 | 56 | 60 | 116
    IC2 or TC2 | 23 | 20 | 43
    IC3 or TC3 | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: The Median Survival Time Will be Determined.
Description: The time from the start of treatment to death
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SBRT Plus Gemcitabine | SBRT Plus Pembrolizumab and Trametinib
Number analyzed (Participants) | 85 | 85
months | 12.8 [11.2 to 14.4] | 14.9 [12.7 to 17.1]

2. Secondary Outcome: One- and Two-year Overall Survival Rate Will be Determined.
Description: The number of patients alive at 1 year and 2 years.
Time Frame: 2 year
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT Plus Gemcitabine | SBRT Plus Pembrolizumab and Trametinib
Number analyzed (Participants) | 85 | 85
Participants
  1-year OS rate | 48 | 53
  2-year OS rate | 0 | 2

3. Secondary Outcome: Treatment-related Adverse Effects Will be Determined.
Description: Treatment-related adverse effects are determined by National Cancer Institute Common Toxicity Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT Plus Gemcitabine | SBRT Plus Pembrolizumab and Trametinib
Number analyzed (Participants) | 85 | 85
Participants
  Grade 3 pyrexia | 0 | 2
  Grade 3 vomitting | 2 | 1
  Grade 3 and 4 increased ALT or AST | 6 | 10
  Grade 3 stomatitis | 0 | 1
  Grade 3 rash | 0 | 2
  Grade 3 and 4 neutropenia | 9 | 1
  Grade 3 thrombocytopenia | 4 | 1
  Grade 3 increased blood bilirubin | 0 | 4
  Grade 3 hypokalemia | 0 | 1
  Grade 3 hyponatremia | 0 | 3
  Grade 3 pneumonia | 0 | 1
  Grade 3 hypertension | 0 | 2

4. Secondary Outcome: The Median Progression Free Survival Time Will be Determined.
Description: The time from the start of treatment until documentation of any clinical or radiological disease progression or death, whichever occurred first. Progression is assessed by the Response Evaluation Criteria in Solid Tumors (RECIST; version 1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SBRT Plus Gemcitabine | SBRT Plus Pembrolizumab and Trametinib
Number analyzed (Participants) | 85 | 85
months | 5.4 [3.2 to 7.6] | 8.2 [6.9 to 9.5]

5. Secondary Outcome: One- and Two-year Progression Survival Rate Will be Determined. Will be Determined.
Description: The proportion of patients without disease progressions at 1 year and 2 years.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT Plus Gemcitabine | SBRT Plus Pembrolizumab and Trametinib
Number analyzed (Participants) | 85 | 85
Participants
  1-year PFS rate | 7 | 18
  2-year PFS rate | 0 | 0

6. Secondary Outcome: The Quality of Life Will be Analyzed.
Description: The analysis of quality of life is based on European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (QLQ-C30). All scales and subscales range from 0 to 100. Regarding physical functioning, role functioning, emotional functioning, cognitive functioning, social functioning and global health, higher scores may indicate better outcomes. In the case of fatigue, nausea and vomitting, pain, dyspnea, insomina, appetite loss, constipation, diarrhea and financial difficulties, lower scores may indicate better outcomes. Scales of all items are independent and not combined to compute a total score.
Time Frame: 3 years
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | SBRT Plus Gemcitabine | SBRT Plus Pembrolizumab and Trametinib
Number analyzed (Participants) | 85 | 85
units on a scale
  Physical functioning | 86.2 [80 to 93.3] | 83.7 [73.3 to 93.3]
  Role functioning | 81.8 [66.7 to 100] | 84.5 [66.7 to 100]
  Emotional functioning | 73.9 [58.3 to 91.7] | 72.1 [58.3 to 83.3]
  Cognitive functioning | 84.7 [66.7 to 100] | 83.3 [66.7 to 100]
  Social functioning | 85.5 [83.3 to 100] | 84.1 [66.7 to 100]
  Global health | 83.6 [75 to 91.7] | 83.2 [75 to 91.7]
  Fatigue | 29.6 [10 to 43.3] | 26.6 [10 to 43.3]
  Nausea and vomitting | 29.4 [16.7 to 50] | 28.8 [0 to 50]
  Pain | 23.9 [0 to 50] | 26.5 [16.7 to 50]
  Dyspnea | 16.1 [0 to 33.3] | 13.7 [0 to 33.3]
  Insomina | 14.9 [0 to 33.3] | 17.6 [0 to 33.3]
  Appetite loss | 31.0 [0 to 66.7] | 33.3 [0 to 66.7]
  Constipation | 14.5 [0 to 33.3] | 16.5 [0 to 33.3]
  Diarrhea | 15.7 [0 to 33.3] | 15.7 [0 to 33.3]
  Financial difficulties | 16.8 [0 to 33.3] | 17.2 [0 to 33.3]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | SBRT Plus Gemcitabine | SBRT Plus Pembrolizumab and Trametinib
All-Cause Mortality (participants affected / at risk) | 85/85 | 83/85
Serious Adverse Events (participants affected / at risk) | 21/85 | 29/85
Other Adverse Events (participants affected / at risk) | 85/85 | 85/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SBRT Plus Gemcitabine (N=85) | SBRT Plus Pembrolizumab and Trametinib (N=85)
Grade 3 pyrexia (General disorders) | 0 | 2
Grade 3 vomitting (Gastrointestinal disorders) | 2 | 1
Grade 3 and 4 increased ALT or AST (Hepatobiliary disorders) | 6 | 10
Grade 3 stomatitis (Gastrointestinal disorders) | 0 | 1
Grade 3 rash (Skin and subcutaneous tissue disorders) | 0 | 2
Grade 3 and 4 neutropenia (Blood and lymphatic system disorders) | 9 | 1
Grade 3 thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1
Grade 3 increased blood bilirubin (Hepatobiliary disorders) | 0 | 4
Grade 3 hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Grade 3 hyponatremia (Metabolism and nutrition disorders) | 0 | 3
Grade 3 pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Grade 3 hypertension (Cardiac disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SBRT Plus Gemcitabine (N=85) | SBRT Plus Pembrolizumab and Trametinib (N=85)
Grade 1-2 Nausea and vomitting (Gastrointestinal disorders) | 17 | 11
Grade 1-2 diarrhea (Gastrointestinal disorders) | 16 | 18
Grade 1-2 increased ALT or AST (Hepatobiliary disorders) | 12 | 16
Grade 1-2 stomatitis (Gastrointestinal disorders) | 0 | 8
Grade 1-2 rash (Skin and subcutaneous tissue disorders) | 2 | 14
Grade 1-2 neutropenia (Blood and lymphatic system disorders) | 21 | 6
Grade 1-2 thrombocytopenia (Blood and lymphatic system disorders) | 15 | 7
Grade 1-2 proteinuria (Renal and urinary disorders) | 2 | 5

LIMITATIONS AND CAVEATS:
The major limitation of the study was the small number of the randomized patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-05): https://cdn.clinicaltrials.gov/large-docs/56/NCT02704156/Prot_SAP_000.pdf